CLINICAL TRIAL: NCT04036084
Title: Développement de Nouveaux Biomarqueurs en Imagerie Par résonance magnétique Pour Les études Longitudinales Dans l'Angiopathie CADASIL
Brief Title: Development of New Biomarkers With Magnetic Resonance Imaging for Longitudinal Studies in CADASIL Angiopathy
Acronym: BIOMRI_CADA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP180325
Record Dates: First submitted 2019-07-15; First posted 2019-07-29 (Actual); Last update posted 2020-08-18 (Actual); Status verified 2020-07

CONDITIONS: Cadasil; Angiopathy; Cerebral
MeSH Terms: conditions — CADASIL

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Patients with CADASIL disease : Diagnosis confirmed by the detection of a pathogenic mutation in the NOTCH3 gene characteristic of CADASIL
  Interventions: Diagnostic Test: Cerebral Magnetic resonance imaging (MRI)
- Control
  Interventions: Diagnostic Test: Cerebral Magnetic resonance imaging (MRI)

INTERVENTIONS:
Diagnostic Test: Cerebral Magnetic resonance imaging (MRI) — Cerebral Magnetic resonance imaging (MRI) 3 Tesla at Inclusion Cerebral Magnetic resonance imaging (MRI) 3 Tesla at Month 1 Cerebral Magnetic resonance imaging (MRI) 3 Tesla at Year 1

SUMMARY:
CADASIL (Cerebral Autosomal Dominant Arteriopathy with Subcortical Infarcts and Leukoencephalopathy) is an cerebral microangiopathy secondary to mutations in the NOTCH3 gene located on chromosome 19. This disease is the most frequent of the hereditary vascular leukoencephalopathies.

CADASIL begins between the ages of 20 and 40 with the appearance of hyper-signs of brain white matter visible on T2 sequences in magnetic resonance imaging (MRI). Before the age of 30, patients are most often asymptomatic. The disease is then responsible for different neurological manifestations:

1. Migraine attacks with aura occur on average in one in three patients, most often at the beginning of the course of the disease, sometimes even before the appearance of MRI abnormalities;
2. Transient ischemic strokes or strokes associated with small cerebral infarcts occur most frequently after the age of 50-60 years in more than two out of three patients;
3. Mood disorders are reported by one in three patients in the same age group;
4. Cognitive disorders that affect executive functions, especially after the age of 60, until the stage of severe dementia associated with walking disorders are observed during the course of the disease.

To date, there is no treatment whose efficacy has been proven in CADASIL. Various studies have shown that the accumulation of the most destructive brain tissue lesions at the subcortical level was closely correlated in CADASIL with the clinical severity of patients (motor and cognitive disability). It is now possible to measure microstructural changes in brain tissue in diffusion imaging during the course of the disease, even before significant clinical changes are detected.

ELIGIBILITY:
Inclusion Criteria:

Patients

* Age from 18 to 80 years
* Confirmed diagnosis (detection of a pathogenic mutation of the NOTCH3 gene)
* Detailed clinical and MRI assessment of the disease (follow-up at the CERVCO) including Rankin score <4
* Any contraindication to MRI or EEG examination (claustrophobia, presence of material with magnetic properties)
* Social security insurance
* Written consent.

Controls

* Age from 18 to 80 years
* No history of neurological or psychiatric diseases
* No history of migraine with aura
* No history of vascular disease (peripheral arteries, heart, brain)
* No known or treated diabetes
* No known or treated hypercholesterolemia
* Social security insurance
* Written consent

Exclusion Criteria:

Patients

* Patients with a contraindication to MRI or EEG examination (claustrophobia, material with magnetic properties: pacemaker, ferromagnetic material ...)
* For MRI examination of neurovascular coupling: Patients with a treatment that may interfere with neurovascular coupling (in particular any treatment with non-steroidal anti-inflammatory drugs, psychotropic drugs, antihypertensive agents or statins)
* Patients without a social security insurance
* Patients under the age of 18 or over 80 at the time of the first visit
* Patients unable to give their informed consent
* Person referred to in Articles L. 1121-5 to L. 1121-8 and L. 1122-12 of the Public Health Code, defined by:

  * Pregnant, parturient or nursing woman
  * Person deprived of liberty by judicial or administrative decision
  * Person hospitalized without consent and not subject to a legal protection measure, and person admitted to a health or social institution for purposes other than research
  * Minor
  * Adult under legal protection measure (guardianship, guardianship or court order), an adult unable to express their consent and not subject to a protective measure
  * Person submitted to an exclusion period for another research (washout period)

Controls

* Subject with a contraindication to MRI or EEG examination (claustrophobia, material with magnetic properties: pacemaker, ferromagnetic material ...)
* For MRI examination of neurovascular coupling: Subject with a treatment that may interfere with neurovascular coupling (in particular any treatment with non-steroidal anti-inflammatory drugs, psychotropic drugs, antihypertensive agents or statins)
* Subject without a social security insurance
* Subject under the age of 18 or over 80 years at the time of the first visit
* Patients unable to give their informed consent
* Person referred to in Articles L. 1121-5 to L. 1121-8 and L. 1122-12 of the Public Health Code, defined by:

  * Pregnant, parturient or nursing woman
  * Person deprived of liberty by judicial or administrative decision
  * Person hospitalized without consent and not subject to a legal protection measure, and person admitted to a health or social institution for purposes other than research
  * Minor
  * Adult under legal protection measure (guardianship, guardianship or court order), an adult unable to express their consent and not subject to a protective measure
  * Person submitted to an exclusion period for another research study (washout period)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CADASIL patients with a proven NOTCH3 mutation
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-08-10 (Actual); Primary Completion 2022-07-06 (Estimated); Study Completion 2023-01-06 (Estimated)

PRIMARY OUTCOMES:
Intra-axonal | 1 year
  Intra-axonal volume fraction
Extra-axonal | 1 year
  Extra-axonal volume fraction
Intra-myelinic edema | 1 year
  Volume fraction of intra-myelinic edema
Microvascular compartment fraction measured using diffusion MRI (IVIM) | 1 year
  Measures of the Flowing blood volume fraction (corresponding to slow intra-voxel incoherent motion (IVIM) of water molecules in the cerebral microvasculature at voxel level)
variation | 1 year
  Overall variation of cerebral blood flow over 20 and 40 seconds stimulations (area under a curve)
blood flow | 1 year
  Maximum cerebral blood flow measured over 20 and 40 seconds stimulations
Slope | 1 year
  Slope of the regression curve when cerebral blood flow is measured 15 and 35 seconds after the onset of the stimulation
Dynamics of the cerebral blood | 1 year
  Dynamics of the cerebral blood flow curve between 15 and 35 seconds (model with dual component responses; fast (before 20 seconds) and slow (after 20 seconds))

CONTACTS AND LOCATIONS:
Locations (1):
- Lariboisiere hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided